CLINICAL TRIAL: NCT03390673
Title: A Phase I, Double-blind, Randomised, Single-dose, Parallel Group Study to Demonstrate the Equivalent Pharmacokinetic Properties of a Single Intravenous Dose of HD204 and Bevacizumab (Avastin®) in Healthy Male Subjects
Brief Title: To Demonstrate Equivalent Pharmacokinetic Properties of HD204 and Bevacizumab (Avastin®) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prestige Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: SAMSON-1
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
Keywords: randomized; double-blind
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HD204 (Experimental): Bevacizumab Single-Dose 1mg/kg body weight by 90 minute intravenous infusion
  Interventions: Drug: HD204
- EU-licensed Avastin (Active Comparator): Bevacizumab Single-Dose 1mg/kg body weight by 90 minute intravenous infusion
  Interventions: Drug: Avastin
- US-licensed Avastin (Active Comparator): Bevacizumab Single-Dose 1mg/kg body weight by 90 minute intravenous infusion
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: HD204 — Single-Dose 1mg/kg body weight by 90 minute intravenous infusion
  Other Names: Bevacizumab
  Arms: HD204
Drug: Avastin — Single-Dose 1mg/kg body weight by 90 minute intravenous infusion
  Other Names: Bevacizumab
  Arms: EU-licensed Avastin; US-licensed Avastin

SUMMARY:
The purpose of this study is to compare the pharmacokinetics, as well as to evaluate the safety, tolerability and immunogenicity of HD204, US-Avastin and EU-Avastin in healthy male subjects after intravenous administration of a single dose..

DETAILED DESCRIPTION:
This is a double-blind, randomized, three-arm, parallel-group, single-dose study. A total of 120 evaluable subjects are required.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking healthy male subjects, 18-50 years old inclusive
* Body Mass index is between 19 to 30 kg/m2, inclusive
* NO history of hypersensitivity or allergic reaction to the active ingredient, murine proteins, or excipients, spontaneous or following drug administration.
* For subjects with female partners of child-bearing potential, an adequate form of contraception must be adhered to prior to entry into the study and for a further 3 months after the end of study. Adequate contraception is defined as the usage by the female partner of any form of hormonal contraception or intra-uterine device (which should be established prior to the start of study) plus usage by one of the partners of an additional spermicide-containing barrier method of contraception. The use of a barrier method alone or reliance on abstinence is not considered adequate.
* Subjects must agree not to donate sperm during the study and for 4 months following treatment with the study medication or until scheduled End Of Study (EOS), whichever is longer.
* Subjects must be able to communicate well with the investigator, to understand and comply with the requirements of the study, and understand and sign the written informed consent.

Exclusion Criteria:

* Clinically significant abnormalities in physical examination, laboratory test results or electrocardiogram (ECG)
* Systolic blood pressure > 140 mmHg or < 90 mmHg , or diastolic blood pressure > 90 mmHg or <50 mmHg
* Proteinuria (with a urine dipstick value of 2+ or above)
* Coagulation abnormalities ( i.e., INR > 2x ULN)
* Bleeding diathesis, history of duodenal ulcers, concomitant use of anticoagulants, or any hemorrhage within 6 months prior to study enrollment.
* Surgical procedure within 2 months of screening, or planned surgical procedure within 2 months of EOS
* Positive test result for drugs of abuse or alcohol breathing test.
* Positive test result for hepatitis B surface antigen (HBsAg), hepatitis C (HCV), or human immunodeficiency virus (HIV) 1 or 2.
* Donated or lost > 500ml of blood in the previous 3 months
* Taken an investigational drug within 3 months (or 5 half-lives), whichever is longer.
* Taken any prescription medications within 14 days or 5 half-lives (whichever is longer) of the first dose of study drug or non-prescription drugs (with the exception of paracetamol, which is allowed).
* Previously received bevacizumab or any product considered to be biosimilar to bevacizumab, or any other antibody or protein targeting VEGF or VEGFR.
* Unwillingness or inability to comply with the study protocol for any reason.
* Male subject whose partner is pregnant.
* History or evidence of a clinically significant disorder (including cardiovascular, cerebrovascular, endocrine or psychiatric), or immunocompromised condition, or disease that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* History of alcohol and/or drug abuse within 12 months of screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Area under Curve (AUC, Pharmacokinetics) | up to week 12
  Sampling will be performed in all patients to compare the PK through values of HD204 and Avastin

SECONDARY OUTCOMES:
Immunogenicity | Days 1 (predose), 15, 22,29, 36, 43, 50, 64, 78 and 95(End of treatment)
  Incidence of anti-bevacizumab antibodies
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) | From Day 1 through study completion (Day 95)
  Safety and tolerability will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events and CTC v4.03

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Christchurch Clinical Studies Trust Ltd, Christchurch

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Demarchi M, Coliat P, Barthelemy P, Schott R, BenAbdelghani M, Kim M, Hii JCS, Feyaerts P, Ang FRX, Derde MP, Deforce F, Petit T, Schwabe C, Wynne C, Park LS, Pivot X. A randomized phase I study comparing the pharmacokinetics of a bevacizumab (HD204) biosimilar to European Union- and United States of America-sourced bevacizumab. PLoS One. 2021 Sep 23;16(9):e0248222. doi: 10.1371/journal.pone.0248222. eCollection 2021. PMID 34555031